CLINICAL TRIAL: NCT02752932
Title: TumorGraft- Guided Therapy for Improved Outcomes in Head and Neck Squamous Cell Cancer- A Feasibility Study
Acronym: Xenograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Champions Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 106515
Record Dates: First submitted 2016-02-24; First posted 2016-04-27 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; Patient derived Xenograft; Chemotherapy; Metastases
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HNSCC -PDX development (Other): Participants with HNSCC who will undergo curative surgery will be included in this group. This involves PDX development only, no drug testing will be done on the PDX.
  Interventions: Other: Drug testing on PDX per Investigator's choice (upto 4)
- RMHNSCC -PDX drug testing (Other): Participants with RMHNSCC who are under palliative treatment will be included in this group. Drug testing on PDX per Investigator's choice (upto 4): PDX will be developed and upto four Chemotherapeutics (that are funded in Ontario) will be tested on the PDX. Chemotherapeutics will be selected at the discretion of the treating Medical Oncologists. Result of the drug testing will be provided to the responsible physician and can be utilized in patient care.
  Interventions: Other: Drug testing on PDX per Investigator's choice (upto 4)

INTERVENTIONS:
Other: Drug testing on PDX per Investigator's choice (upto 4) — Drug of Investigator's choice (upto 4 Ontario funded Chemotherapeutics) will be tested on PDX (Patient Derived Xenografts)

SUMMARY:
Primary objectives:

1. Evaluate the feasibility of rapidly accruing 30 participants with recurrent metastatic head and neck squamous cell carcinoma for the development of patient derived xenographs (PDX) from fresh, real time biopsies in which sensitivity to < 4 Ontario funded chemotherapeutic regimen will be tested. Written feedback to the primary oncologist will be provided.
2. There is also a curative intent cohort of 30 participants undergoing surgical resection with curative intent. These PDX models will undergo exome sequencing with written feedback.
3. Feasibility in both surgical and recurrent cohorts will be a measure of i) engraftment rate, ii) patient status at the time of drug testing completion and iii) rate of accrual.

DETAILED DESCRIPTION:
Tumour samples from 30 participants with HNSCC that undergone curative surgery will be used to establish patient-derived xenografts (PDXs). These tumours will also undergo exome sequencing. This will provide a biobank of PDX models with available genomic information for future research projects. Another 30 participants with recurrent or metastatic HNSCC (RMHNSCC) will be recruited to this study. PDX models will be developed from these patient tumours, followed by genomic sequencing. PDX models are developed by transplanting small tumour pieces into immunocompromised mice. These mice are then treated with different available drugs for RMHNSCC at the discretion of their medical oncologist. These mice will be then followed up to examine the tumour response to treatments. When studied in clinic, PDX models have shown high correlation with patient response to the treatment. The PDX drug testing results will be provided to the treating medical oncologist to guide care at the oncologists discretion. Investigators' hope is that improved chemotherapy responses are observed with this strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent metastatic squamous cell carcinoma of the head and neck.
2. Lesion amenable to biopsy (1 cm or more)
3. Lesion capable of yielding 4 biopsy cores
4. 18 years or older
5. Capable of providing and signing for informed consent

Exclusion Criteria:

1. Cognitive impairment prohibitive to providing informed consent
2. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
To determine the rate of PDX engraftment for HNSCC and RMHNSCC samples | 1-2 years
Time to engraftment | 1-2 years
Percentage of models successfully undergoing drug testing | 1-2 years
Participant status at the time of completion of drug testing | 1-2 years
  Participant status at the time of completion of drug testings(i.e. what percentage of participants are alive and well enough to receive further chemo).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Nichols, MD, FRCSC, Principal Investigator — London Regional Cancer Program; Eric Winquist, MD, FRCPC, Principal Investigator — London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided